CLINICAL TRIAL: NCT05502380
Title: Broad-spectrum Antibiotic Prophylaxis in Tumor and Infected Orthopedic Sur-gery - the Prospective-randomized, Microbiologist-blinded, Stratified, Superiority Trials - BAPTIST Trials
Brief Title: Broad-spectrum Antibiotic Prophylaxis in Tumor and Infected Orthopedic Surgery
Acronym: BAPTIST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BASEC 2022-00800
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Surgical Site Infection; Microbial Colonization; Antibiotic Resistant Infection
Keywords: Perioperative antibiotic prophylaxis; Selection; High Risk patients; Ranndomized-Controlled Trial
MeSH Terms: conditions — Surgical Wound Infection; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: At enrollment (Day 1), the investigator will prescribe the preoperative antibiotic prophylaxis based on instructions provided in the protocol according to the patient's randomization. Patients will be randomized in the ratio 1:1 into the investigational group (broad-spectrum prophylaxis) and the control group (usual prophylaxis). Each patient can be included several times with one episode for each surgical interven-tion in the operating theatre. The initial consent form is valid during 1 month and will be renewed in case of another inclusion following a delay of 1 month after the initial signature of the patient.
Who Masked: Care Provider
Masking Description: The microbiologists culturing the pathogens of eventual surgical site infections are blinded to the prior prophylaxis during the index surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard prophylaxis arm (Active Comparator): The standard prophylaxis consists of one to three intravenous doses of cefuroxime 1.5 g intravenously; or cefuroxim 3g if obesity > 120 kg or a BMI > 35 kg/m2; or vancomycin 1 g or clindamycin 600 mg in case of intolerance to cephalosporins
  In patients alrady under current therapuetic antibiotic therapy, continuation of that therapuetic antibiotic regimen
  Interventions: Drug: Standard antibiotic prophylaxis
- Innovative prophylaxis arm (Experimental): Additional single-shot perioperative antibiotic prophylaxis with Broad-spectrum prophylaxis: vancomycin 1 g & gentamicin 5 mg/kg.
  Interventions: Drug: Standard antibiotic prophylaxis

INTERVENTIONS:
Drug: Standard antibiotic prophylaxis — One to three intravenous doses of cefuroxime 1.5 g intravenously; or 3g if obesity; or vancomycin 1 g or clindamycin 600 mg; if allergy. Continuation of eventual current therapeutic antibiotc regimens for any infection

SUMMARY:
The perioperative antibiotic prophylaxis is evidence-based in orthopedic surgery. While its duration ranges from a single dose to three doses throughout the world, the choice of the prophylactic agents is undisputed. Worldwide, the surgeons use 1st or 2nd-generation cephalosporins (or vancomycin in some cases).

However, there are particular clinical situation with a high risk of antibiotic-resistant surgical site infections (SSI); independently of the duration of adminis-tered prophylaxis. These resistant SSI's occur in contaminated wounds, or during surgery under current therapeutic antibiotics, and base on "selection" by antibiotics used for therapy or for prophylaxis.

DETAILED DESCRIPTION:
The perioperative antibiotic prophylaxis is evidence-based for the majority of orthopedic surgeries. While the debate of its duration and timing (single-dose versus triple-dose; before or after the intraoperative microbiological sampling) may continue, no clinicians doubt on the efficiency of the recommended prophylactic agents; that are mostly 1st or 2nd-generation cephalosporins, co-amoxiclav or other exceptional agents in cases of (pseudo)-allergy. However. and traditionally, up to the half of all detected pathogens of orthopedic SSI's are not covered by the prior prophylactic regimens: e.g. SSIs due to methicillin-resistant cocci or non-fermenting Gram-negative rods in orthopedic surgery.

Additionally, orthopedic surgeons operating selected patient populations (neoplasms, open fractures, postoperative wound dehiscence9, diabetic foot infections or already infected body sites) experience a high risk of prophylactic-resistant pathogens, or pathogens resistant to current therapeutic antibiotics regimens. At least 10% of all new intraoperative tissue samples, during iterative surgical debridement, yield (new) pathogens unknown to the clinicians.

This is due to selection by prophylactic or therapeutic antibiotics, which only kill the previously detected pathogens, but left over newly introduced contaminants, remnant parts of partially-diagnosed polymicrobial infections; ultimately leading to a new SSIs occurring during therapy for the first infection at the orthopedic site. This selection is unpredictable involving both Gram-positive skin pathogens as well as (multi) resistant Gram-negative rods.From a microbiological point of view, only a maximal Gram-negative coverage, alongside with a large Gram-negative coverage, would cover these selections.

The literature is in-existing how to prevent these selections. Most clinicians just continue with the standard prophylactic recommendation, or the current thera-peutic antibiotic regimen. Theoretically, clinicians cannot exclude that these selected patient populations eventually might profit from a broad-spectrum prophylaxis.

The BAPTIST trials only concern the perioperative antibiotic prophylaxis in selected situations of orthopedic surgery: tumor surgery, debridement for postoperative dehiscent wounds, debridement under antibiotics, open fractures, skin colonization with multidrug-resistant bacteria, plus, as a control; spine surgery in selected multimorbid patients. The investigators alternately randomize the standard prophylaxis (or by continuing the current antibiotic treatment) to the additional broad-spectrum single-shot of vancomycin 1g IV & single-shot of gentamicin 5 mg/kg intravenously; before an eventual intraoperative sampling. End-of-Treatment (EOT) and/or Test-of-Cure (TOC) occur latest at the 6-week's surgical control visit. The rest of the hospital stay, treatment, the use of negative-pressure vacuum therapy, other interventions, local antibiotic therapies; therapies or procedure are at the discretion of the treating clinicians.

The investogators will randomize surgical interventions defined by the inclusion criteria in a prospective-alternating scheme (1:1) according to the scheduled position in the operating theatres. The anesthetists (or the nurses at the hospitalization units) the will administer the standard prophylaxis (or the therapeutic antibiotics) alone, or with the addition of the single-shot broad-spectrum prophylaxis regimen composed of vancomycin and gentamicin. In case of clinical suspicion of infection or massive contamination, the surgeons will perform at least three microbiological intraoperative tissue samples. Each surgery counts as an independent event. If a patient is debrided several times, he/she can have different prophylaxis regimens during each of the interventions. After the prophylactic regimen, the clinicians are free to continue with a targeted or empirical therapeutic antibiotic regimen. The antibiotic therapy per se is not an objective of this current trials.

The treatment period includes the following daily study visits:

* Visit 1 - Enrollment (Day 1)
* EOT (end of microbiological cultures) - Day 14 (+/- 3 days)
* TOC (clinical surgical control) - Day 42 (+/- 14 days)
* Follow-up (telephone) for implant-related surgery - 1 year (+/- 2 months)

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Surgery under current or recent therapeutic antibiotics (antibiotic-free window <14 days and past antibiotic prescription >4 days)
* Surgery for open fractures and wounds; including 2nd and 3rd looks
* Potentially contaminated wound revision in the operating theatre
* Tumor (oncologic) surgery (if prior radiotherapy and/or bone involvement)
* Spine surgery with ASA-Score >= 3 points, sacral involvement, or re-vision surgery
* Known skin colonization with multidrug-resistant Gram-negative bacteria

Exclusion Criteria:

* Inability to understand the study procedure for linguistic or cognitive rea-sons
* Surgery without intraoperative microbiological samples
* Allergy or major intolerance to vancomycin and/or gentamicin
* Anticipated clinical follow-up of less than 6 weeks after inclusion
* Pregnant or breastfeeding women
* Known carriage of multiresistant Gram-negative bacteria in the urine or anal region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infections (SSI) at 6 weeks for surgeries without implant; and 1 year for surgeries with implant | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  Assessment of SSI at the clinical controls according to clinical criteria in the literature (pus, discharge, pain, inflammation, several deep tissue microbiological cultures

SECONDARY OUTCOMES:
Proportion of antibiotic-resistant pathogens in the deep surgical site of the study patients; in relation to the prior antibiotic prophylaxis or the current therapeu-tic antibiotic therapy | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  Assessments of antibiotic resistance of pathogens according to standard susceptibilty testing in the Microbiological Laboratory
Incidence of revision surgery for non-infections reasons within 6 weeks | 6 weeks postoperatively
  Unplanned revision surgery in the operating theatre for any reasons
Proportion of the change of antibiotic therapy based on intraoperative findings | 6 weeks postoperatively
  Asssesment in the medical files. Have therapeutic antibiotics been changed according to new intraoperative bacterial culture findings
Incidence of dverse events and global costs of therapeutic antibiotics (if any) | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  If there is therapeutic antibiotc treatment necessary, the investigators assess the drugs, the adverse events and the global costs related to the antibiotc treatment. The costs are the global (overall) hospitalizations costs in Swiss Francs.
Incidence of non-SSI infections within 6 weeks (e.g. urine infections) | 6 weeks postoperatively
  Assessment of all nosocomial and community-acquired infections ocrruging in the immediate postoperative period and relate them to prior perioperative antibiotic prophylaxis
Incidence of skin and body colonization with Gram-negative multi-resistant bacteriaweeks (if there are any samples) | 4-6 weeks postoperatively
  Assessment of the impact of the priorantibiotic prophylaxis on the body colonization with multiresistant bacteria of concern for infection control

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, Professor, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators might share anonomyzed key elements (data) upon scientific request to the corresponding person
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2025
Access Criteria: The ivestigators might bilaterally share anonomyzed key elements (data) upon scientific request to the corresponding person

REFERENCES:
- [Background] Uckay I, Hoffmeyer P, Lew D, Pittet D. Prevention of surgical site infections in orthopaedic surgery and bone trauma: state-of-the-art update. J Hosp Infect. 2013 May;84(1):5-12. doi: 10.1016/j.jhin.2012.12.014. Epub 2013 Feb 14. PMID 23414705
- [Background] Wuarin L, Abbas M, Harbarth S, Waibel F, Holy D, Burkhard J, Uckay I. Changing perioperative prophylaxis during antibiotic therapy and iterative debridement for orthopedic infections? PLoS One. 2019 Dec 18;14(12):e0226674. doi: 10.1371/journal.pone.0226674. eCollection 2019. PMID 31851708
- [Background] Jamei O, Gjoni S, Zenelaj B, Kressmann B, Belaieff W, Hannouche D, Uckay I. Which Orthopaedic Patients Are Infected with Gram-negative Non-fermenting Rods? J Bone Jt Infect. 2017 Jan 15;2(2):73-76. doi: 10.7150/jbji.17171. eCollection 2017. PMID 28529866
- [Background] Muller D, Kaiser D, Sairanen K, Studhalter T, Uckay I. Antimicrobial Prophylaxis for the Prevention of Surgical Site Infections in Orthopaedic Oncology - A Narrative Review of Current Concepts. J Bone Jt Infect. 2019 Oct 15;4(6):254-263. doi: 10.7150/jbji.39050. eCollection 2019. PMID 31966954
- [Derived] Uckay I, Bomberg H, Risch M, Muller D, Betz M, Farshad M. Broad-spectrum antibiotic prophylaxis in tumor and infected orthopedic surgery-the prospective-randomized, microbiologist-blinded, stratified, superiority trials: BAPTIST Trials. Trials. 2024 Jan 19;25(1):69. doi: 10.1186/s13063-023-07605-5. PMID 38243311